CLINICAL TRIAL: NCT03107065
Title: A Pilot, Open-Label, Single-Center, Single-Treatment, Safety And Effectiveness Evaluation Of Percutaneous-Temperature Controlled-Radiofrequency Electrocoagulation Used To Contract Tissue Associated With Axillary Sweat Glands
Brief Title: Single-Treatment, Study of Percutaneous-Temperature Controlled-RF Electrocoagulation on Axilla Tissue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ThermiGen, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: THERMI_0007
Record Dates: First submitted 2016-12-08; First posted 2017-04-11 (Actual); Last update posted 2017-12-20 (Actual); Status verified 2017-12

CONDITIONS: Sweating Increased Armpits
Keywords: Sweating

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- single treatment (Experimental): Percutaneous-Temperature Controlled-Radiofrequency Electrocoagulation Used To Contract Tissue Associated With Axillary Sweat Glands
  Interventions: Device: Thermi Radiofrequency

INTERVENTIONS:
Device: Thermi Radiofrequency — Percutaneous-Temperature Controlled-Radiofrequency Electrocoagulation

SUMMARY:
This is a pilot, open-label, and single-center, single-treatment prospective evaluation of the electrocoagulation of axillary sweat gland tissue using the ThermiRF device to improve excessive sweating of the axilla(s).

In this study, "Temporary Relief" is defined as improvement on the DLQI.

Twenty male and female subjects between 18 and 50 years old will be enrolled. A total of five visits are planned for this study.

A punch biopsy will be collected (prior to and post treatment and analyzed to determine the degree of impact to the tissue after the electrocoagulation treatment.

Safety assessments will be collected using the Numerical Rating Scale (NRS) a 10-point scale, and adverse events reports (observed or reported).

The total length of the study is approximately 4 months.

DETAILED DESCRIPTION:
This is a pilot, open-label, and single-center, single-treatment prospective evaluation of the electrocoagulation of axillary sweat gland tissue using the ThermiRF device to alleviate or improve symptoms associated with axillary sweating.

In this study, "Temporary Relief" is defined as improvement on the DLQI.

A total of 20 male and female healthy volunteers between the age of 18 and 50 will be enrolled in this study. Subjects who sign the informed consent form and meet all entry criteria will be assigned a unique number/code to preserve confidentiality.

A total of five visits are planned for this study as described below:

* Visit 1: Screening visit - (Day 0)
* Visit 2: Single Treatment
* Visit 3: Day 30 (± 7 days)
* Visit 4: Day 60 (± 7 days)
* Visit 5: Day 90 (± 7 days)

A punch biopsy will be collected at Visit 1(screening), Visit 2 (post-treatment) and Visit 4 (Day 60). The purpose of the punch biopsy is to evaluate the degree of impact to the axillary organ after the electrocoagulation treatment when compared to pre-treatment at Visit 1.

Safety assessments will be collected using the Numerical Rating Scale (NRS) a 10-point scale, and adverse events reports (observed or reported).

The total length of the study is approximately 4 months.

ELIGIBILITY:
5Inclusion Criteria

* Male or female between the age of 18 and 50 inclusive
* Focal, visible excess sweating present for at least 6 months
* Self-reported excess sweating that becomes visible through clothing and has a negative psychosocial impact on the subject's quality of life
* At least any two of the following:

  * Bilateral and symmetrical excessive sweating
  * Impairs activities of daily life
  * At least one episode per week
  * Age of onset <25 years
* Desire to reduce / improve the condition
* Willing to refrain the use of deodorant products containing "Aluminum Chloride" one to two weeks prior to treatment and for the duration of the study
* Females of childbearing potential who are sexually active must be willing to use an approved method of birth control during study participation
* Cooperative, reliable, and able to read and comprehend English
* Able to read, understand, sign and date the informed consent document (English only)
* Able and willing to comply with the schedule visit(s) and study requirements.

Exclusion Criteria

Subjects presenting with any of the following will not be included in the study

* Prior use of botulinum toxin injections into axilla within the last 6 months
* Priory Miradry treatments
* Prior surgical dissection, curettage or liposuction
* Current or prior sympathectomy
* Current or prior laser therapy to axilla for hyperhidrosis
* Female subject in menopause stage
* Current use of oral medications such as oxybutynin, glycopyrolate, clonazepam, clonidine, phenoxybenzamine or propranolol
* Use within 7 days preceding surgery of ibuprofen, , non-steroidal anti-inflammatory products, or any products including herbals and supplements that could interfere with the clinical assessments of this study (other than drugs used for anesthesia)
* Subjects who have a pacemaker, implantable defibrillators, metal stents, implants or other monitoring equipment
* History or current injury to the axilla or nearby anatomical areas.
* Clinically significant wounds, lesions or acute infections including, dermatitis, lupus or other autoimmune disease affecting the dermis
* Pregnant or planning pregnancy prior to the end of study participation
* History or current diagnosis of cancer of any type
* History of uncontrolled cardiovascular disease(i.e. myocardial infarction, hypertension, hypercholesterolemia, peripheral vascular disease)
* Known hypersensitivity to local anesthetic medications
* History, or current bleeding disorders (i.e. hemophilia or von Willebrand disease), or anticipated treatment with prescription anticoagulants
* History of AIDs/HIV
* Serious mental health illness such as dementia or schizophrenia; psychiatric hospitalization in the past two years
* Developmental disability or cognitive impairment that would preclude adequate comprehension of the informed consent form and/or ability to follow study subject requirement and/or record the necessary study measurements
* Any family member of the investigator or investigational staff, or an employee of the investigator.
* Participation in any other investigational study within 30 days prior to consent;

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-12-08 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-09-06 (Actual)

PRIMARY OUTCOMES:
Dermatology Life Quality Index (DLQI) improvement post treatment | Day 60
  subjective improvement from initial to post questionnaire on the DLQI

OTHER OUTCOMES:
Odor Scale (OS) Improvement post treatment | Day 60 and Day 90
  subjective improvement from initial to post questionnaire on the OS
Reduction of excessive sweating | Day 60
  Reduction of 1-point improvement on the HDSS

CONTACTS AND LOCATIONS:
Overall Officials: Toni Fournier, Study Director — ThermiGen, LLC; Kevin O'Brien, Study Chair — ThermiGen, LLC
Locations (1):
- Faces+ Plastic Surgery, Dermatology, Skin and Laser, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No